CLINICAL TRIAL: NCT04658368
Title: Patient Reported Outcomes Following Targeted Muscle Reinnervation in Major Limb Amputees
Brief Title: Patient Reported Outcomes Following Targeted Muscle Reinnervation
Status: Terminated | Type: Observational
Why Stopped: After research hold, study never restarted and was subsequently terminated.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1466; A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison); Protocol Version 11/2020 (Other: UW Madison)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Amputation
Keywords: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Participants with a history of major limb amputation at the University of Wisconsin (UW) that did not undergo TMR
- Retrospective TMR: Participants with a history of major limb amputation that underwent primary or secondary TMR with attending plastic surgeon at UW
  Interventions: Procedure: Primary TMR; Procedure: Secondary TMR
- Prospective Secondary TMR: Participants who are scheduled to undergo secondary TMR at the UW
  Interventions: Procedure: Secondary TMR
- Prospective Primary TMR: Participants who are scheduled to undergo primary TMR at the UW
  Interventions: Procedure: Primary TMR

INTERVENTIONS:
Procedure: Primary TMR — TMR procedure as part of the primary major limb amputation surgery
  Groups: Prospective Primary TMR; Retrospective TMR
Procedure: Secondary TMR — TMR procedure subsequent to major limb amputation surgery
  Groups: Prospective Secondary TMR; Retrospective TMR

SUMMARY:
The purpose of this study is to characterize the functional status and quality of life of patients undergoing Targeted Muscle Reinnervation (TMR) at time of major limb amputation (primary) or subsequent to major limb amputation (secondary). Participants can expect to be on study for about a year and will complete a short electronic survey and option phone interview.

DETAILED DESCRIPTION:
Residual limb pain and phantom limb pain (PLP) have been shown to be associated with decrease in prosthetic function and poor quality of life. It is estimated that the prevalence of PLP is as high as 85% and residual limb pain 10-76%. The treatment of amputee-related pain continues to rely largely on pharmacologic therapy, and typically opioids. Targeted Muscle Innervation (TMR) first performed by Dr. Dumanian, is a peripheral nerve transfer procedure that reroutes amputated axons to motor endplates and sensory organelles in nearby muscles, giving amputated nerves "somewhere to go and something to do" which may play a role in preventing development of neuromas and phantom limb pain.

A multicenter retrospective study found that upper-extremity amputees who subsequently underwent TMR ("secondary TMR") experienced relief in neuroma pain post-operatively. Other studies have shown that amputees who have undergone TMR have decreased narcotic use and improvement in prosthetic tolerance. A randomized controlled trial demonstrated that major limb amputees who underwent TMR had decreased phantom limb pain and residual limb pain compared with those who underwent traditional treatment of neuroma excision and burying into muscle. A subsequent study found that patients undergoing major limb amputation with immediate TMR ("primary TMR") had less PLP and residual limb pain than untreated amputee controls. A recent prospective study of patients undergoing TMR at time of major limb amputation secondary to trauma had overall low pain scores, and neuromodulator medication use and overall high rate of daily prosthetic use. Oncologic patients who underwent amputation with concurrent TMR demonstrated decreased neuroma symptoms, PLP and residual limb pain compared to oncologic amputees who did not undergo TMR. However, 32% of patients who underwent TMR for upper extremity amputation did not finish prosthetic rehabilitation, despite showing overall improved functional outcome scores.

Thus, there is increasing evidence that TMR, both primary and secondary, can prevent or improve pain from neuroma, phantom and residual limb pain. There is also evidence that TMR may promote early use of prosthetics and reduce reliance on narcotic medications. Prior studies have largely relied on outcome measures such as Numerical Rating Scale (NRS) for pain and pain-related instruments from the Patient-Reported Outcomes Measurement Information System (PROMIS) toolbox. More comprehensive data is limited on patient's functional status and quality of life, and thus far there is a lack of studies using patient-reported outcome instruments specific to patients with upper or lower extremity conditions. There is also limited data on patient desires and expectations for pursuing TMR, and subsequent satisfaction after having undergone the procedure.

Retrospective Cross-sectional study: Medical record review, electronic survey, optional interview This is a mixed methods, cross-sectional study assessing major limb amputee patients who have undergone TMR. It includes a medical record review to collect demographic information listed below, and an electronic survey (quantitative study), as well as interviews with a subset of subjects (qualitative study). Patients who have had at least 6 months follow up will be invited to participate in the electronic survey, which will include questions from validated patient-reported outcome instruments to measure function and quality of life. Patients will also be invited to be interviewed by phone using a set of open-ended questions. Thematic content analysis will be used to evaluate the participants' responses, and with the objective to examine the patient's motivations for undergoing TMR and their postoperative course, including pain, daily function, quality of life.

Prospective Cohort study: Medical record review, electronic survey, optional interview This is a mixed methods cohort study of patients with history of major limb amputation who will be undergoing secondary TMR, and patients who will be undergoing a major limb amputation with primary TMR. It includes a medical record review to collect demographic information listed below. The pre-survey will be administered between time of pre-operative evaluation to just prior to the operation, and the post-survey will be administered between 6-18 months after surgery. Each subject will also be invited to be interviewed by phone (or in person if at University of Wisconsin for follow up appointment), with set of open-ended questions focused on motivations for undergoing TMR, and their postoperative course including pain, daily function, quality of life.

General amputee population: Electronic survey ONLY To define normative data for general amputee population, the electronic survey with patient reported outcomes measures will be administered to amputees recruited from prosthetic, orthotic, orthopedic, vascular, oncologic or other amputee clinics and support groups.

For all above, the electronic survey, which will be administered via REDCap, will take approximately 7-8 minutes to complete. The interview will take 15-20 minutes to complete.

Study Aims:

* Aim 1: Evaluate functional status and quality of life of patients who have undergone primary or secondary TMR using patient reported outcome instruments
* Aim 2: Compare functional status and quality of life of primary TMR patients to those of general amputee population
* Aim 3: Compare pre-operative and post-operative functional status and quality of life of secondary TMR patients
* Aim 4: Compare post-operative functional status and quality of life of secondary TMR patients to those of general amputee population
* Aim 5: Evaluate patient desire, expectations and satisfaction with undergoing TMR (via survey and structured interview)

ELIGIBILITY:
Inclusion Criteria: Study cohort

* Retrospective

  * Underwent primary or secondary TMR with attending plastic surgeon at UW
* Prospective

  * Patient with history of major limb amputation who is scheduled to undergo secondary TMR with attending plastic surgeon at UW
  * Patient who is scheduled to undergo primary major limb amputation with concurrent TMR

Inclusion Criteria: Control Cohort

* Patient with history of major limb amputation recruited from local clinics who has not been referred or seen for consultation for TMR by attending plastic surgeon at UW

Exclusion Criteria: Study Cohort

* Retrospective

  * Patient underwent TMR at another institution
  * Less than 6 months follow up
  * Less than 18 years of age
  * Enrolled in other studies relating to neuropathic pain
  * Undergoing radiation therapy
  * Incarcerated
  * Incomplete survey response
  * Non-English speaking (chosen PROMIS measures only in English)
* Prospective

  * Less than 18 years of age
  * Cognitive impairment
  * Enrolled in other studies relating to neuropathic pain
  * Undergoing radiation therapy
  * Incarcerated
  * Non-English speaking (chosen PROMIS measures only in English)

Exclusion Criteria: Control Cohort

* Less than 18 years of age
* Cognitive impairment
* Enrolled in other studies relating to neuropathic pain
* Undergoing radiation therapy
* Incarcerated
* Incomplete survey response
* Major limb amputee seeking consultation for TMR
* Non-English speaking (chosen PROMIS measures only in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone (retrospective) or are scheduled to undergo (prospective) major limb amputation with primary or secondary TMR procedure at the UW. A control group of participants that have had major limb amputation at the UW without the TMR procedure will also be surveyed.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Post-Amputation Quality of Life Survey | up to 18 months
  The functional status and quality of life of patients who have undergone primary or secondary TMR will be measured using patient reported outcome instruments. 25-items scored on a 5 point likert scale will be combined for a score between 25 and 125, where higher scores indicate better quality of life. Items represent combined tools of the following PROMIS instruments: Ability to participate in social roles and activities, Global health, Pain intensity, self-efficacy for management chronic conditions social interactions, general self-efficacy, emotional support, social isolation. Higher scores mean better functioning.
Change in Quality of Life Survey | Baseline, post-surgery (up to 18 months)
  Compare pre-operative and post-operative functional status and quality of life of secondary TMR patients. 25-items scored on a 5 point likert scale will be combined for a score between 25 and 125, where higher scores indicate better quality of life. See attachments for more details.
Qualitative Participant TMR Experience | up to 18 months
  Patient desire, expectations and satisfaction with undergoing TMR will be measured qualitatively using survey and semi-structured interview responses. This measure will be analyzed with coding for recurring themes and reported narratively. A coding theme will be decided after preliminary review of interview transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Brett F Michelotti, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No